CLINICAL TRIAL: NCT00075686
Title: A Phase III Randomized Open-Label Study Comparing Gemcitabine Plus Cetuximab (IMC-C225) Versus Gemcitabine As First-Line Therapy Of Patients With Advanced Pancreas Cancer
Brief Title: S0205 Gemcitabine w/ or w/o Cetuximab as First-Line Therapy in Locally Advanced Pancreas Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000347414; S0205 (Other: SWOG); CALGB-S0205 (Other: CALGB); CAN-NCIC-PAC1 (Other: NCIC-CTG); U10CA032102 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine hydrochloride + IMC-C225 (Experimental): Loading dose: gemcitabine hydrochloride 1000mg/m2, IV on Day 1; Cetuxiumab 400mg/m2, IV on Day 1 (cycle 1 only) Weekly maintenance: Cetuximab 250mg/m2, IV on Days 8,15,22 of cycle 1 & days 1,8,15,22 of all subsequent cycles; gemcitabine hydrochloride 1000mg/m2, IV on Days 8,15,22 of cycle 1 and Days 1,8,15 of all subsequent cycles.
  Interventions: Biological: cetuximab; Drug: gemcitabine hydrochloride
- gemcitabine hydrochloride alone (Experimental): gemcitabine hydrochloride 1000mg/m2, IV on Days 1,8,15,22 of cycle 1 and Days 1,8,15 of all subsequent cycles.
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: cetuximab — Loading dose: Cetuxiumab 400mg/m2, IV on Day 1 (cycle 1 only). Weekly maintenance: Cetuximab 250mg/m2, IV on Days 8,15,22 of cycle 1 & days 1,8,15,22 of all subsequent cycles
  Arms: gemcitabine hydrochloride + IMC-C225
Drug: gemcitabine hydrochloride — 1000mg/m2 IV over 30 minutes

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as cetuximab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether gemcitabine is more effective with or without cetuximab in treating pancreatic cancer.

PURPOSE: This randomized phase III trial is studying giving gemcitabine together with cetuximab to see how well it works compared to giving gemcitabine alone as first-line therapy in treating patients with locally advanced unresectable or metastatic adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with locally advanced unresectable or metastatic adenocarcinoma of the pancreas treated with gemcitabine and cetuximab vs gemcitabine alone.
* Compare the time to treatment failure in patients treated with these regimens.
* Estimate the percentage of patients with epidermal growth factor receptor (EGFR) tumor expression in patients treated with these regimens.
* Compare the overall survival of patients in the EGFR-positive subset treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the total response rate (confirmed and unconfirmed complete and partial response) in patients with measurable disease treated with these regimens.
* Compare the patient report of pain and quality of life of patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to disease status (locally advanced unresectable vs metastatic), Zubrod performance status (0 or 1 vs 2), and prior pancreatectomy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, and 22 and gemcitabine IV over 30 minutes on days 1, 8, 15, and 22 for course 1 and days 1, 8, and 15 for all subsequent courses.
* Arm II: Patients receive gemcitabine as in arm I. In both arms, courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each course, and at the end of study therapy.

Patients are followed every 6 months for 2 years and then annually for 1 year.

PROJECTED ACCRUAL: A total of 704 patients (352 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically confirmed pancreatic adenocarcinoma meeting 1 of the following criteria:

  * Locally advanced unresectable disease
  * Distant metastatic disease NOTE: If diagnosis is based on a metastatic site the histology must be compatible with pancreatic cancer
* Measurable or nonmeasurable disease by x-ray, scan, or physical examination
* Tumor tissue must be submitted for evaluation of epidermal growth factor receptor expression before study entry
* None of the following tumor types are allowed:

  * Endocrine tumors
  * Lymphoma of the pancreas
  * Ampullary cancer
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No significant history of cardiac disease
* No uncontrolled hypertension
* No unstable angina
* No uncontrolled arrhythmia
* No congestive heart failure

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer that is currently in remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for advanced pancreatic cancer
* No prior cetuximab or other therapy that targets the epidermal growth factor pathway
* No prior chimerized or murine monoclonal antibody therapy
* No other concurrent anticancer immunotherapy

Chemotherapy

* At least 6 months since prior adjuvant chemotherapy
* No prior chemotherapy or chemoradiotherapy for advanced pancreatic cancer
* No prior gemcitabine
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No prior hormonal therapy for advanced pancreatic cancer
* No concurrent anticancer hormonal therapy

Radiotherapy

* See Chemotherapy
* At least 28 days since prior radiotherapy and recovered
* Prior palliative radiotherapy to metastatic sites allowed
* No concurrent anticancer radiotherapy, including whole brain radiotherapy for progressive disease (i.e., CNS metastasis)

Surgery

* At least 14 days since prior pancreatic cancer surgery and recovered

Other

* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2004-01; Primary Completion 2007-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall survival comparison between treatment groups | every 4 weeks for 3 years

SECONDARY OUTCOMES:
Response rate comparison between treatment groups as measured by RECIST and radiological evaluation at every other course | every 9 weeks until progression
Time to treatment failure comparison between groups from registration to first observation of progressive disease, symptomatic deterioration, or death | every 4 weeks while on treatment
Percentage of patients with EGFR tumor expression and compare overall survival of patients in the EGFR subset | every 4 weeks for 3 years
Toxicity profile comparison of patients treated with 2 regimens and measured until 30 days after completion of study treatment | every 4 weeks while on treatment
Total response rate comparison between treatment groups in the subset of patients with measurable disease by RECIST at every other course | every 9 weeks until progression
Pain and quality of life comparison between treatment groups as measured by patient questionnaire at baseline, before each course, and then completion of study treatment | every 4 weeks while on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute; Eileen O'Reilly, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Ralph PW Wong, MD, FRCPC, Study Chair — CancerCare Manitoba
Locations (389):
- United States (382):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - East Alabama Medical Center, Opelika, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Cancer Center at Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Valley Care Medical Center, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Sutter Solano Medical Center, Vallejo, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Ruby L. Golleher Cancer Program at Presbyterian Intercommunity Hospital, Whittier, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Medical and Surgical Specialists, L L C, Galesburg, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology & Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, P.C. - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Cancer Care at Our Lady of Bellefonte Hospital, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Cancer Treatment Center at Christus Schumpert St. Mary Place, Shreveport, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Mercy Hospital, Portland, Maine
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Cancer Center of Boston - Chestnut Hill, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Hospital, Pontiac, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Kessler Air Force Base, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Health Systems, Kearney, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Seacoast Cancer Center at Wentworth-Douglass Hospital, Dover, New Hampshire
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - San Juan Regional Cancer Center, Farmington, New Mexico
  - New York Oncology Hematology, PC - Albany, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - New York Oncology Hematology, P.C., Latham, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - St. Joseph's Hospital Health Center - Syracuse, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - University Hospitals Ireland Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Huron Hospital Cancer Care Center, Cleveland, Ohio
  - Euclid Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital Cancer Care Center, Warrensville Heights, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, P.C. at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Center for Cancer Medicine and Blood Disorders, PA, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital Regional Cancer Center, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - United Hospital Center, Clarksburg, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center - Elkhorn, Elkhorn, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Medical Center, Racine, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (7):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital of Barrie, Barrie, Ontario
  - Trillium Health Centre - Mississauga Site, Mississauga, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Philip PA, Benedetti J, Fenoglio-Preiser C, et al.: Phase III study of gemcitabine [G] plus cetuximab [C] versus gemcitabine in patients [pts] with locally advanced or metastatic pancreatic adenocarcinoma [PC]: SWOG S0205 study. [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA4509, 2007.
- [Derived] Philip PA, Benedetti J, Corless CL, Wong R, O'Reilly EM, Flynn PJ, Rowland KM, Atkins JN, Mirtsching BC, Rivkin SE, Khorana AA, Goldman B, Fenoglio-Preiser CM, Abbruzzese JL, Blanke CD. Phase III study comparing gemcitabine plus cetuximab versus gemcitabine in patients with advanced pancreatic adenocarcinoma: Southwest Oncology Group-directed intergroup trial S0205. J Clin Oncol. 2010 Aug 1;28(22):3605-10. doi: 10.1200/JCO.2009.25.7550. Epub 2010 Jul 6. PMID 20606093